CLINICAL TRIAL: NCT03086252
Title: Patient-Driven Transfusion Thresholds in Hematological Disorders: A Pilot Study
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow accrual
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Ana G. Antun, MD, Principal Investigator, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00090306; NCI-2016-01059 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); Winship3145-16 (Other: Emory University/Winship Cancer Institute)
Record Dates: First submitted 2017-03-17; First posted 2017-03-22 (Actual); Last update posted 2018-07-26 (Actual); Status verified 2018-07

CONDITIONS: Anemia; Aplastic Anemia; Bone Marrow Failure; Hematopoietic and Lymphoid Cell Neoplasm; Leukemia; Myelodysplastic Syndrome
MeSH Terms: conditions — Anemia; Anemia, Aplastic; Bone Marrow Failure Disorders; Hematologic Neoplasms; Leukemia; Myelodysplastic Syndromes | interventions — Erythrocyte Transfusion; Blood Component Transfusion; Blood Transfusion

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Supportive care (patient-driven RBCT) (Experimental): Patients undergo red blood cell transfusions (RBCT) based on their perception and/or the presence of anemia symptoms for up to 6 months.
  Interventions: Procedure: Red Blood Cell Transfusions (RBCT)

INTERVENTIONS:
Procedure: Red Blood Cell Transfusions (RBCT) — Undergo patient-driven RBCT
  Other Names: Blood Component Transfusion; Blood Transfusion; Transfusion; Transfusion of Blood Products

SUMMARY:
This pilot study evaluates safety of administration of red blood cell transfusions requested by patients based on their symptoms instead of levels of hemoglobin for the treatment of chronic anemia in patients with blood disorders.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To assess feasibility and safety of red blood cell transfusions at the time subjects requested based on symptomatic anemia.

SECONDARY OBJECTIVES:

I. To define a patient-driven red blood cell transfusion (RBCT) threshold and to compare the median hemoglobin (hgb) at the time subjects request RBCT to the standard threshold of hgb < 8 g/dL.

II. To compare the number of red blood cell (RBC) units transfused and the frequency of transfusions at the time subjects request RBCT during the study period to the number of RBC units received and frequency using the standard threshold hemoglobin < 8 g/dL during a comparable period prior to enrollment.

III. To compare the quality of life (QoL) scores when subjects request RBCT to the scores obtained at the time hgb is 8 +/- 0.5 g/dL.

OUTLINE:

Patients undergo RBCT based on their perception and/or the presence of anemia symptoms for up to 6 months.

After completion of study treatment, patients are followed up for 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with hematological malignancy or marrow failure syndrome such as but not limited to: aplastic anemia, myelodysplastic syndrome or leukemia
* Chronic transfusion-dependent anemia with exposure to at least 5 RBCT
* Interested in reducing transfusion exposure
* Willing to sign informed consent

Exclusion Criteria:

* Recent acute bleeding requiring intervention in less than 24 hours
* Hemoglobin levels < 6 g/dL
* Acute leukemia receiving induction chemotherapy
* Any patient with known ischemic heart disease, history of congestive heart failure, history of stroke, or cardiac arrhythmia for which the patient requires medication or a medical device
* Oxygen dependent
* Oxygen saturation below 92% on room air
* Receiving erythropoietin stimulating agent
* Thalassemia major or sickle cell disease requiring blood transfusion
* Undergoing major surgery
* Hemolytic anemia
* Coagulopathies including disseminated intravascular coagulation (DIC), receiving anticoagulant or antiplatelet agents
* Diagnosed with chronic obstructive pulmonary disease (COPD) oxygen dependent
* Pregnancy
* Participation in a therapeutic clinical trial

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-07-24 (Actual); Primary Completion 2018-05-31 (Actual); Study Completion 2018-05-31 (Actual)

PRIMARY OUTCOMES:
Incidence of laboratory and clinical adverse events (AEs) assessed by the Common Terminology Criteria for Adverse Events version 4.03. | Up to 6 months of study participation
  Frequency, duration, and severity of AEs and severe adverse events will be determined. The proportion of subjects with serious side effects will be calculated with 95% confidence interval. Descriptive statistics will be used to characterize subjects enrolled on the trial: age, sex, race and diagnosis.

SECONDARY OUTCOMES:
Frequency of RBC units transfused | Up to 6 months of study participation
  The frequency of RBC units transfused will be compared between study period and prior to enrollment for the same patient (e.g. each patient will serve his/her own control) by Wilcoxon's sign rank test.
Hemoglobin concentration at the time subject requests RBCT | Up to 6 months of study participation
  Hemoglobin concentration (Hgb) will be measured in g/dL.
Number of RBC units transfused | Up to 6 months of study participation
  The number of RBC units transfused will be compared between study period and prior to enrollment for the same patient (e.g. each patient will serve his/her own control) by Wilcoxon's sign rank test.
QoL scores from the Functional Assessment of Cancer Therapy - Anemia/Fatigue (FACT-An) questionnaire at the time hemoglobin is 8 +/- 0.5 g/dL | Up to 6 months of study participation
  Will be compared to QoL scores at the time subjects request RBCT by paired t-test and/or Wilcoxon sign rank test.
QoL scores from the Functional Assessment of Cancer Therapy - Anemia/Fatigue (FACT-An) questionnaire at the time subjects request RBCT | Up to 6 months of study participation
  Will be compared to QoL scores at the time hgb is 8 +/- 0.5 g/dL by paired t-test and/or Wilcoxon sign rank test.

CONTACTS AND LOCATIONS:
Overall Officials: Ana Antun, MD, Principal Investigator — Emory University
Locations (1):
- Emory University/Winship Cancer Institute, Atlanta, Georgia, United States